CLINICAL TRIAL: NCT06076525
Title: Understanding Motor Flexibility and Reactive Balance Control to Improve Fall Prevention Strategies in Older Adults
Brief Title: Motor Flexibility in Multidirectional Balance Control
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol not submitted to IRB
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UNebraska
Record Dates: First submitted 2023-10-01; First posted 2023-10-11 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Falling

STUDY DESIGN:
Intervention Model Description: This is a Parallel Assignment interventional study aimed at investigating the role of behavioral flexibility in multidirectional balance control and fall prevention across different age groups and fall histories. The study will recruit 42 participants divided into three groups: 14 Older Adult Fallers, 14 Older Adult Non-Fallers, and 14 Younger Adult Non-Fallers. Participants will undergo treadmill walking sessions where perturbations in different directions and magnitudes will be introduced. Older Adult Non-Fallers and Younger Adult Non-Fallers will partake in two different aims, involving walking sessions and training epochs. Due to concerns over fatigue, Older Adult Fallers will only participate in one of these aims. The study aims to provide insight into the trade-offs between speed and flexibility in reactive balance control, and the potential for improving balance through targeted interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Older Adult Fallers (participate in Aim 1 only) (Experimental): This group is exposed to the perturbations during treadmill walking in Aim 1 to collect data on their balance control mechanisms.
  Interventions: Behavioral: Multidirectional Perturbations for Balance Control Assessment (60 perturbations)
- Older Adult Non-Fallers - Control Group (participate in Aims 1 and 2) (Active Comparator): This group acts as a comparison for the Older Adult Non-Fallers - Experimental Group within the same demographic.
  Interventions: Behavioral: Multidirectional Perturbations for Balance Control Assessment (60 perturbations)
- Older Adult Non-Fallers - Experimental Group (participate in Aims 1 and 2) (Experimental): This group is exposed to the interventions in both Aims 1 and 2, the latter of which involves targeted training designed to improve their balance control flexibility.
  Interventions: Behavioral: Multidirectional Perturbations for Balance Control Assessment (60 perturbations); Behavioral: Multidirectional Perturbations for Balance Control Assessment (150 perturbations)
- Younger Adult Non-Fallers - Control Group (participate in Aims 1 and 2) (Active Comparator): This group serves as the control for the Younger Adult Non-Fallers - Experimental Group.
  Interventions: Behavioral: Multidirectional Perturbations for Balance Control Assessment (60 perturbations)
- Younger Adult Non-Fallers - Experimental Group (participate in Aims 1 and 2) (Experimental): This group is exposed to the interventions in both Aims 1 and 2, the latter of which involves targeted training designed to improve their balance control flexibility.
  Interventions: Behavioral: Multidirectional Perturbations for Balance Control Assessment (60 perturbations); Behavioral: Multidirectional Perturbations for Balance Control Assessment (150 perturbations)

INTERVENTIONS:
Behavioral: Multidirectional Perturbations for Balance Control Assessment (60 perturbations) — The intervention involves exposing participants to a series of 60 controlled multidirectional perturbations while walking on a treadmill. These perturbations are delivered in varying directions and magnitudes to simulate real-world conditions that might lead to a loss of balance, such as slips or trips. Participants will undergo this series during multiple experimental sessions referred to as epochs. The complete intervention consists of a treadmill familiarization period followed by 5 epochs to assess motor flexibility. Each epoch is followed by a rest period to ensure participant safety and minimize fatigue.
Behavioral: Multidirectional Perturbations for Balance Control Assessment (150 perturbations) — The intervention involves exposing participants to a series of 150 controlled multidirectional perturbations while walking on a treadmill. These perturbations are delivered in varying directions and magnitudes to simulate real-world conditions that might lead to a loss of balance, such as slips or trips. Participants will undergo this series during multiple experimental sessions referred to as epochs. The complete intervention consists of a treadmill familiarization period followed by seven epochs. The first five epochs will deliver multidirectional perturbations to assess modifiability of motor flexibility, followed by a sixth epoch to test generalization to novel perturbation directions while walking. Finally there will be a seventh epoch of perturbations while standing to test generalization from walking balance control to standing balance control. Each epoch is followed by a rest period to ensure participant safety and minimize fatigue.
  Arms: Older Adult Non-Fallers - Experimental Group (participate in Aims 1 and 2); Younger Adult Non-Fallers - Experimental Group (participate in Aims 1 and 2)

SUMMARY:
The goal of this observational study is to learn about how older adults (those 65 and above) manage to maintain balance when experiencing a slip or trip while walking. The study is especially interested in how quickly and flexibly adjustments to movement can be made to avoid falling. The main questions this study aims to answer are:

* How does the ability to adjust movements quickly, also known as "motor flexibility," affect the chances of recovering from a slip or trip?
* Can targeted training improve this ability in older adults, making falls less likely? Participants will walk on a specially designed treadmill that can simulate slips and trips and undergo a training program designed to improve the ability to adjust movements quickly.

Researchers will compare older adults to younger adults to see if age affects the ability to adjust movements quickly and recover balance after a slip or trip. Researcher's will also compare the performance of older adults before and after the training program to see if balance recovery improves.

DETAILED DESCRIPTION:
Falls are the leading cause of injury-related fatalities in people aged 65 and above, often triggered by unexpected disruptions like slips or trips during walking. Such events necessitate rapid and adaptable motor responses to regain balance, a mechanism referred to as "reactive balance control." Within this complex interplay, "motor flexibility," or the ability to modulate one's movements in real-time based on sensory feedback, becomes critical. However, there exists a trade-off: increased flexibility requires more complex sensory processing, potentially delaying the initiation of corrective actions-a delay that can prove perilous in the context of a fall. This study seeks to explore the role of motor flexibility in reactive balance control, particularly in older adults, with a focus on understanding how individuals adapt stepping patterns in response to diverse and unpredictable balance disturbances. State-of-the-art technology will be employed including a Computer-Assisted Rehabilitation Environment (CAREN), to simulate various types of walking surface disruptions. By studying younger and older adults and introducing different types of perturbations, the study aims to understand the trade-offs between the speed of motor response and the flexibility to adapt to different fall scenarios. Additionally, the extent to which training can improve this balance control flexibility is investigated. The central hypothesis is that motor flexibility is a modifiable feature of reactive balance control and is positively correlated with the ability to recover from multi-directional disturbances. The study will quantify this relationship and assess the potential for improvement through targeted interventions. Aim 1 of the research is designed to measure these trade-offs in older adults by introducing controlled perturbations to a walking platform, thereby providing critical data on how speed and flexibility interact in real-world fall scenarios. Computational models will be used to evaluate how these variables contribute to an individual's ability to resist falls from varying directions and magnitudes. Aim 2 will explore the potential for improving balance control flexibility through targeted training, studying both younger and older adults to gauge the effects of age on the adaptability of motor control. Improvements in balance flexibility and determine how these changes interact with other physiological factors like body mass index and rate of force development. The results of this study will provide foundational data that can be used to develop more effective fall-prevention strategies for older adults. This research bridges biomechanics and computational modeling, offering an interdisciplinary lens through which to view a problem of substantial public health significance. By understanding the nuances of how motor flexibility and reaction speed interact in the context of unexpected balance disturbances, we aim to make strides in mitigating the risks and consequences of falls in older adults.

ELIGIBILITY:
Inclusion Criteria:

* The proposed study will include individuals from two distinct age ranges, between 19 to 35 years old and 65 to 79 years old. This approach ensures a wide demographic representation and allows for comparison across different age groups.

Exclusion Criteria:

* Uncontrolled hypertension
* Peripheral arterial disease
* Knee osteoarthritis
* Vertigo
* Meniere's disease
* Chronic dizziness
* History of back or lower extremity injury that currently limits completing multidirectional perturbation protocol
* Prior surgery that affects the subject's mobility
* Any neurological disease or impairment that limits the ability to walk, including but not limited to stroke, Parkinson's disease, and multiple sclerosis.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Motor Flexibility Index in Reactive Balance Control | Immediately after intervention
  The Motor Flexibility Index is quantified using the coefficient of determination (R-squared) from a linear regression model that predicts recovery step placement based on the multi-directional motion state of the upper body 100 milliseconds after disturbance onset. A higher R-squared value indicates better motor flexibility, reflecting an individual's ability to adaptively respond to unexpected balance disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel H Hunt, PhD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie the results reported in publications arising from this study will be shared, including demographic data, behavioral assessments, and outcomes. This will also encompass data dictionaries to enable future researchers to understand the variables used. No sensitive identification information will be included in the shared dataset to protect participant privacy.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The IPD will become available starting 6 months after the publication of summary data and will remain accessible for a period of 5 years thereafter. This is to provide adequate time for the research team to fully analyze and publish initial findings, and to ensure that the IPD remains relevant and useful to the research community.
Access Criteria: Access to IPD will be granted to qualified researchers for the purposes of conducting secondary analyses. Requests for IPD should be submitted to the principal investigator.